CLINICAL TRIAL: NCT05306080
Title: Pilot, Open-Label Study Evaluating the Safety and Feasibility of Using Rescue Therapies for CAR T Cell Related Cytokine Release Syndrome (CRS) and HLH-like Syndrome
Brief Title: Tadekinig Alfa (IL-18BP) Rescue Therapy for CAR T Cell Related Cytokine Release Syndrome (CRS) and HLH-like Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01422
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: CRS - Cytokine Release Syndrome; HLH
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — interleukin-18 binding protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tadekinig alfa (Experimental): * Injection #1/Day 1: As clinically indicated in accordance with Figure 1.1-1.
  * Repeat Injection(s): Missed doses will not be made up.
  * Injection #2/Day 3: Approximately 48 hours (+/- 5 hours) after receipt of the 1st injection.
  * Injection #3/Day 5: Approximately 48 hours (+/- 5 hours) after receipt of the 2nd injection.
  * Continued Dosing (Optional): Approximately q48-72 hours; If the subject is responsive to initial therapy, but has ongoing symptoms of CRS/CRHLS.
  * Retreatment (Optional): May be considered
  Interventions: Drug: Tadekinig alfa (IL-18BP)

INTERVENTIONS:
Drug: Tadekinig alfa (IL-18BP) — Tadekinig alfa will be administered via subcutaneous injection. The site of subcutaneous injection should be rotated to avoid injection site reactions; e.g. the outside of the thighs, arms, and the various quadrants of the anterior abdominal wall.
  * Injection #1/Day 1:
    o Loading dose of 4 mg/kg; Maximum dose of 350 mg.
  * Repeat Injection(s): 2 mg/kg/injection; Maximum dose of 160 mg/injection. Missed doses will not be made up.
    * Injection #2/Day 3: Approximately 48 hours (+/- 5 hours) after receipt of the 1st injection.
    * Injection #3/Day 5: Approximately 48 hours (+/- 5 hours) after receipt of the 2nd injection.
    * Continued Dosing (Optional): Approximately q48-72 hours; If the subject is responsive to initial therapy, but has ongoing symptoms of CRS/CRHLS.

SUMMARY:
This is a pilot, open-label study to assess the safety and feasibility of using investigational drug(s) as rescue therapies for CAR T cell related CRS and HLH-like syndrome (CRHLS).

DETAILED DESCRIPTION:
This pilot, open-label trial will allow for co-enrollment of subjects participating in University of Pennsylvania-Sponsored, CCI-Initiated CAR T cell studies. As utilization of this investigational drug may be required emergently in the event of qualifying safety events post CAR T cell infusion, subjects may be consented/enrolled at the time they receive an investigational CAR T cell product. If/when use of this investigational drug is deemed clinically necessary, rescue therapy may then be initiated.

Cohort 1: Will allow for the use of Tadekinig alfa, an interleukin-18 binding protein that binds and neutralizes IL-18. IL-18 is a key mediator in systemic inflammatory conditions such as MAS/HLH, which may contribute to the severity of CAR T cell-related cytokine release syndrome (CRS) and HLH-like syndrome (CRHLS) and impact response to standard therapy. In addition, subjects experiencing other IL-18 driven toxicity post CAR T cell therapy which is non-responsive to conventional treatment may also receive rescue therapy with Tadekinig alfa as per clinical discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written informed consent
2. Male or female patients age ≥ 18 years
3. Have been co-enrolled in a University of Pennsylvania-Sponsored, CCI-Initiated CAR T cell clinical trial.
4. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in protocol

Exclusion Criteria:

1. Pregnant or nursing (lactating) women.
2. Known hypersensitivity to the active substance or one of the excipients of the investigational product(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate preliminary safety and feasibility of administering investigational rescue therapies for the treatment of CAR T cell related CRS and CRHLS. | 28 days
  Type, frequency, and severity of AEs/SAEs determined to be related to the rescue therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided